CLINICAL TRIAL: NCT03948191
Title: A Double-masked, Methylprednisolone-control, Efficacy and Safety Study of 99Tc-MDP for Thyroid Associated Ophthalmopathy.
Brief Title: 99Tc-MDP for Thyroid-Associated Ophthalmopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dalian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: zsyy_nfm2-2017-10
Record Dates: First submitted 2019-05-10; First posted 2019-05-13 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Thyroid-Associated Ophthalmopathy
Keywords: 99Tc-MDP; TAO; efficacy; safety
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylprednisolone(ivMP) (Active Comparator): Methylprednisolone(ivMP) 500mg i.v. infusion once a week for 6 weeks followed by 250mg i.v. once a week for 6 weeks.
  Interventions: Drug: Methylprednisolone
- 99Tc-MDP (Experimental): 99Tc-MDP 15mg i.v. infusion once a day for 10 days, 20 days apart, received 3 courses of infusions.
  Interventions: Drug: 99Tc-MDP(99Technetium-Methylenediphosphonate Injection)

INTERVENTIONS:
Drug: Methylprednisolone — 500mg i.v. infusion once a week for 6 weeks followed by 250mg i.v. once a week for 6 weeks.
  Arms: Methylprednisolone(ivMP)
Drug: 99Tc-MDP(99Technetium-Methylenediphosphonate Injection) — 15mg i.v. infusion once a day for 10 days, 20 days apart, received 3 courses of infusions.
  Other Names: Yunke
  Arms: 99Tc-MDP

SUMMARY:
To investigate the efficacy，safety and tolerability of 99Tc-MDP in comparison to Methylprednisolone, in the treatment of participants suffering from active moderate to severe TAO.

ELIGIBILITY:
Inclusion Criteria:

* The patient age 18 Years to 76 Years;
* Fewer than 6 months from onset of TAO;
* Clinical diagnosis of Graves' disease associated with active TAO and a clinical activity score of ≥ 3;
* Moderate to severe TAO;
* No previous medical or surgical treatment, excluding local supportive measures and oral steroids if the maximum cumulative dose is less than 1000 mg methylprednisolone or equivalent with at least 6 weeks between last administration of oral steroids and randomization.

Exclusion Criteria:

* Optic neuropathy, severe orbital appearance and surgical;
* Extra-thyroid disease;
* Pregnant and children;
* Severe impairment of cardiac, hepatic and renal functions;
* Allergies;
* Other contraindications.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Responder Status at Week 12 | Week 12
  This end point main evaluation improvement of clinical activity score and proptosis at week 12. A reduction of the CAS 2 point or more, and reduction of the proptosis 2 mm or more was defined as response.

SECONDARY OUTCOMES:
Overall Average Continuous Change in CAS From Baseline to Week 24 | Baseline to Week 24
  The 7-item European Group on Graves' Ophthalmopathy (EUGOGO) amended CAS was used to evaluate clinical activity. CAS of 3 point or more on a 7-point scale indicating active thyroid-associated ophthalmopathy.
Overall Average Continuous Change in Proptosis From Baseline to Week 24 | Baseline to Week 24
  Proptosis is the amount of protrusion of the eye from the orbital rim. Measurements were recorded with the Hertel exophthalmometer.
Overall Average Change in Diplopia grading From Baseline to Week 24 | Baseline to Week 24
  Diplopia grading included 01/4no：no diplopia; 11/4intermittent： diplopia in primary position of gaze, when tired or when first awakening; 21/4inconstant： diplopia at extremes of gaze; 31/4constant： continuous diplopia in primary or reading position).
  Diplopia change in one grade or more at week 24 was regarded as improvement.
Overall Average Change in extra-ocular muscular thickening From Baseline in thickening extra-ocular muscular improvement in Orbital CT to Week 24 | Baseline to Week 24
  Observation of extra-ocular muscular thickening is observed on Orbital CT. One or more extra-ocular muscle recovery at week 24 was regarded as improvemed.
Overall Average Change in Graves' Ophthalmopathy Quality of Life (GO-QOL) Scale From baseline to Week 24 follow-up | Baseline to Week 24
  The GO-QOL is a 16-item self-administered questionnaire used to assess the perceived effects of thyroid associated ophthalmopathy (TAO) by the participants on their daily physical and psychosocial functioning. Two subscales of the 16-question GO-QOL have been defined: Visual Functioning and Appearance, with 8 questions comprising each subscale.The transformed overall score is the sum of scores from all 16 questions to a scale of 0 (worst health) to 100 (best health). A change of 8 point was defined as improvement.
Overall Average Change in GO-QOLScale - Visual Functioning From baseline to Week 24 follow-up | Baseline to Week 24
  Transformed Visual Functioning score is the sum of scores from following 8 questions to a scale of 0 (worst health) to 50 (best health): bicycling, driving, moving around the house, walking outdoors, reading, watching television (TV), hobby or pastime, feel hindered.
Overall Average Change in GO-QOLScale - Appearance From baseline to Week 24 follow-up | Baseline to Week 24
  Transformed Appearance score is the sum of scores from the following 8 questions to a scale of 0 (worst health) to 50 (best health): feel appearance has changed, feel being stared at, feel people react unpleasantly, influence on self-confidence, feel socially isolated, influence on making friends, appear less often on photos, try to mask changes in appearance.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided